CLINICAL TRIAL: NCT00166517
Title: Immunogenicity and Safety of V260 in Healthy Infants in Korea
Brief Title: V260 Registration Study (V260-013)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V260-013; 2005_071
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Results first posted 2009-09-23 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Rotavirus
Keywords: Gastrointestinal Rotavirus
MeSH Terms: interventions — Rotavirus Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): RotaTeq
  Interventions: Biological: Rotavirus Vaccine, Live, Oral, Pentavalent
- 2 (Placebo Comparator): Placebo
  Interventions: Biological: Comparator: Placebo

INTERVENTIONS:
Biological: Rotavirus Vaccine, Live, Oral, Pentavalent — 3 doses of rotavirus vaccine live, oral, pentavalent on Day 1, 28 to 70 days post Dose 1, and 28 to 70 days post Dose 2
  Arms: 1
Biological: Comparator: Placebo — 3 doses of placebo to rotavirus vaccine live, oral, pentavalent on Day 1, 28 to 70 days post Dose 1, and 28 to 70 days post Dose 2
  Arms: 2

SUMMARY:
Immunogenicity and Safety of V260 in Healthy Infants in Korea

ELIGIBILITY:
Inclusion Criteria:

* At first study vaccination, age 6 weeks through exactly 12 weeks

Exclusion Criteria:

* History of congenital abdominal disorders, intussusception, or abdominal surgery
* History of known prior rotavirus disease
* Ongoing chronic diarrhea or failure to thrive
* Clinical evidence of active gastrointestinal illness

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 178 (Actual)
Dates: Start 2005-08; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Kim DS, Lee TJ, Kang JH, Kim JH, Lee JH, Ma SH, Kim SY, Kim HM, Shin SM. Immunogenicity and safety of a pentavalent human-bovine (WC3) reassortant rotavirus vaccine in healthy infants in Korea. Pediatr Infect Dis J. 2008 Feb;27(2):177-8. doi: 10.1097/INF.0b013e31815aba79. PMID 18174862

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 8 sites.in Korea from 02-Aug-2005 (first patient in) to 25-May-2006 (last dose
  given). Last subject completed follow-up: 05-Jul-2006. All data corrections applied (Frozen File) on 18-
  Aug-2006
Pre-assignment Details: Subjects with history of congenital abdominal disorders, intussusception, or abdominal surgery; history of
  known prior rotavirus disease; ongoing chronic diarrhea or failure to thrive and those with clinical evidence
  of active gastrointestinal illness were excluded.
Groups:
- RotaTeq™: Three oral doses of RotaTeq™ (rotavirus vaccine, live, oral, pentavalent) administered 28 to 70 days apart, with up to 42 days of safety follow-up after each vaccination.
- Placebo: Placebo matching RotaTeq™ administered 28 to 70 days apart, with up to 42 days of safety follow-up after each vaccination.
Period: Overall Study
Arm/Group | RotaTeq™ | Placebo
Started | 115 | 63
Vaccinated at Visit 1 | 115 | 63
Vaccinated at Visit 2 | 112 | 61
Vaccinated at Visit 3 | 110 | 61
Completed | 110 | 61
Not Completed | 5 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 4 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RotaTeq™ | Placebo | Total
Number analyzed (Participants) | 115 | 63 | 178
Age, Customized [Number; unit: participants]
  6-12 Weeks of Age | 114 | 63 | 177
  Over 12 Weeks of Age | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 30 | 76
  Male | 69 | 33 | 102

OUTCOME MEASURES:

1. Primary Outcome: Serum Anti-Rotavirus IgA Response
Description: Number of subjects with ≥ 3-fold rise from baseline (Predose 1) in
  Serum IgA 14 days Postdose 3
Time Frame: Baseline and 14 days Postdose 3
Population: Per Protocol Population
Measure: Number; unit: Participants
Arm/Group | RotaTeq™ | Placebo
Number analyzed (Participants) | 94 | 52
Participants | 89 | 7
Statistical Analysis 1: Comparison: RotaTeq™; Test type: Non-Inferiority or Equivalence — Non-inferiority was assessed versus a constant, 85%, based on historical data; p = 0.003, Exact test of proportion — p ≥.85, where p is the proportion of subjects who achieved ≥3-fold rise from baseline in the group that received RotaTeq®; Exact test of proportion, based on binomial distribution

2. Secondary Outcome: Serum Neutralizing Antibody (SNA) Response to Serotypes G1, G2, G3, G4 and P1A
Description: Number of subjects with ≥ 3-fold rise from baseline (Predose 1) in
  SNA response to G1, G2, G3, G4 and P1A 14 days Postdose 3
Time Frame: Baseline and 14 days Postdose 3
Population: Per Protocol Population
Measure: Number; unit: Participants
Arm/Group | RotaTeq™ | Placebo
Number analyzed (Participants) | 94 | 52
Participants
  Number of subjects with ≥ 3-fold rise in SNA to G1 | 67 | 2
  Number of subjects with ≥ 3-fold rise in SNA to G2 | 34 | 1
  Number of subjects with ≥ 3-fold rise in SNA to G3 | 42 | 1
  Number of subjects with ≥ 3-fold rise in SNA to G4 | 62 | 4
  Number of subjects with ≥3-fold rise in SNA to P1A | 65 | 3

ADVERSE EVENTS:
Time Frame: Patients in this study were followed for all adverse experiences, for 42 days following each study vaccination.
Description: The number of patients listed in the Adverse Event tables (RotaTeq™ and Placebo) is the number of patients who received study treatment.
  Although a patient may have had two or more clinical adverse experiences the patient is counted only once in a category. The same patient may appear in different categories.
Arm/Group | RotaTeq™ | Placebo
Serious Adverse Events (participants affected / at risk) | 6/114 | 7/63
Other Adverse Events (participants affected / at risk) | 110/114 | 63/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RotaTeq™ (N=114) | Placebo (N=63)
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Acute bronchiolitis (Infections and infestations) | 0 | 1
Bronchiolitis (Infections and infestations) | 3 | 0
Bronchitis (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 3 | 1
Otitis media acute (Infections and infestations) | 1 | 2
Pneumonia (Infections and infestations) | 0 | 1
Pneumonia mycoplasmal (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Burn (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RotaTeq™ (N=114) | Placebo (N=63)
Acute tonsillopharyngitis (Blood and lymphatic system disorders) | 1 | 0
Acute tonsillopharyngitis mild (Blood and lymphatic system disorders) | 0 | 1
Laryngomalacia (Congenital, familial and genetic disorders) | 1 | 0
Conjunctival injection (Eye disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 2 | 2
Eye discharge (Eye disorders) | 6 | 1
Eye disorders (Eye disorders) | 1 | 0
Strabismus (Eye disorders) | 0 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 5 | 4
Diarrhoea (Gastrointestinal disorders) | 59 | 34
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Loose stools (Gastrointestinal disorders) | 2 | 3
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 65 | 33
Fever (General disorders) | 25 | 17
Irritability (General disorders) | 97 | 52
Atopy (Immune system disorders) | 3 | 2
Acute bronchiolitis (Infections and infestations) | 1 | 1
Acute pharyngitis (Infections and infestations) | 4 | 5
Bronchiolitis (Infections and infestations) | 13 | 5
Bronchitis (Infections and infestations) | 12 | 3
Chickenpox (Infections and infestations) | 1 | 0
Cold (Infections and infestations) | 10 | 4
Croup (Infections and infestations) | 2 | 0
Enteritis (Infections and infestations) | 1 | 0
Enterovirus infection (Infections and infestations) | 1 | 0
Folliculitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 13 | 4
Impetigo (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 3 | 0
Otitis externa (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 4 | 1
Otitis media acute (Infections and infestations) | 4 | 1
Perianal abscess (Infections and infestations) | 2 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 3 | 1
Rhinitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 44 | 36
Urinary tract infection (Infections and infestations) | 1 | 0
Scratch (Injury, poisoning and procedural complications) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Oral intake reduced (Metabolism and nutrition disorders) | 1 | 1
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Fear (Psychiatric disorders) | 2 | 0
Food aversion (Psychiatric disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal stuffiness (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 9 | 6
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 1
Diaper rash (Skin and subcutaneous tissue disorders) | 2 | 2
Facial rash (Skin and subcutaneous tissue disorders) | 0 | 1
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 1
Skin rash (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0
Vesicle (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.